CLINICAL TRIAL: NCT04338958
Title: A Phase-II Clinical Trial for First Line Treatment of Stage II/III Covid-19 Patients to Treat Hyperinflammation
Brief Title: Ruxolitinib in Covid-19 Patients With Defined Hyperinflammation
Acronym: RuxCoFlam
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas Hochhaus, Principal Investigator, University of Jena
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RuxCoFlam
Record Dates: First submitted 2020-04-07; First posted 2020-04-08 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19 | interventions — ruxolitinib

STUDY DESIGN:
Intervention Model Description: single arm, non-randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib (Experimental): 2 x 10mg Ruxolitinib with defined response adapted dose escalation up to 2 x 20mg for a duration of 7 days
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — 2 x 10mg Ruxolitinib with defined response adapted dose escalation up to 2 x 20mg for a duration of 7 days with clinical and/or radiographic response assessment

SUMMARY:
RuxCoFlam is a single arm, non-randomized open phase II trial for front line treatment of Covid-19 patients with defined hyperinflammation.

DETAILED DESCRIPTION:
RuxCoFlam is a single arm, non-randomized open phase II trial for front line treatment of Covid-19 patients with defined hyperinflammation. Purpose of the study is the reversal of hyperinflammation to improve pulmonary function, reduce respiratory dependency and reduce mortality. Patients with a hyperinflammation Score 10/16 without a clinical diagnosis of sepsis will be treated with 2 x 10mg Ruxolitinib with defined response adapted dose escalation up to 2 x 20mg for a duration of 7 days with clinical and/or radiographic response assessment. Inflammation assessment will be performed every other day (day 3, 5,7) using the CIS. In patients with unaffected CIS alteration < 25% or increasing CIS > 25% dose escalation by 5mg steps (15mg, day3; 20mg day 5) at the investigator´s discretion. Treatment can be extended up to 28 days if clinically indicated and the benefits of treatment outweigh the risks. Primary endpoint of the study is the overall response rate in reversal of hyperinflammation at day 7 compared to baseline. Secondary endpoints are total use of assisted oxygenation dependency (duration (days) of invasive/non-invasive ventilation or duration (days) of high-flow Oxygen support), radiologic response (reversal of pulmonary Covid-signs, Lung-XRay/CT), day 15 clinical status and day 15 and day 29 mortality. Patients aged ≥18 years hospitalized with COVID-19 pneumonia (demonstrated by CXRAY or chest CT), with a study specific Covid Inflammation Score ≥ 10 are eligible. Patients with active tuberculosis or uncontrolled bacterial, fungal, viral, or other infection (besides SARS-CoV-2 virus) will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient or guardian must provide written informed consent (and assent if applicable) before any study assessment is performed.
* 2. Male and female patients aged ≥ 18 years.
* 3. Patients with temperature > 37.3°C
* 4. Patients with respiratory symptoms and/or hypoxia SpO2 < 93%
* 5. Patients with Covid-19 stage II and stage III
* 6. Patients with lung imaging showing bi-pulmonary infiltrates (chest X-ray or CT scan).
* 7. Patients, with a Covid Inflammation Score ≥ 10

Exclusion Criteria:

* 1. History of hypersensitivity to any drugs or metabolites of similar chemical classes as ruxolitinib.
* 2. Uncontrolled active bacterial, fungal, viral, or other infection (besides COVID-19).
* 3. Active Tuberculosis infection.
* 4. Known Positivity for HBV, HCV or HIV.
* 5. Patients who are on long-term use of oral anti-rejection or immunomodulatory drugs
* 6. Participating in any other interventional clinical trial for COVID-19.
* 7. Treatment with cytokine-directed agents such as anti-IL6 or anti-IL1R directed antibodies (i.e. tocilizumab, anakinra). Other treatment modalities used in locally adapted SOPs (corticosteroids, chloroquine, hydroxychloroquine, lopinavir-ritonavir) may be given with daily documentation of dose and schedule.
* 8. ALT or AST > 5 x ULN detected within 24 hours at screening (according to local laboratory reference ranges).
* 9. ANC < 500/µL at screening (according to local laboratory reference ranges).
* 10. Platelet count < 50,000/µL at screening (according to local laboratory reference ranges).
* 11. Hemoglobin < 6 g/dl (3.73mmol/l)
* 12. Pregnant or nursing (lactating) women.
* 13. Female patients of childbearing potential (e.g. are menstruating) and male patients who do not agree to abstinence or, if sexually active, do not agree to the use of highly effective contraception as defined below, throughout the study and for up to 90 days after stopping treatment, OR Female patients of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception as defined below, throughout the study and for up to 90 days after stopping treatment.

Highly effective contraception methods include:

* Total abstinence (when this is in line with the preferred and usual lifestyle of the patient). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
* Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that patient.
* Use of oral, injected or implanted hormonal methods of contraception. Placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception (in case of oral contraception, patients should have been using the same pill on a stable dose for a minimum of 3 months before Screening).

Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
overall response rate in reversal of hyperinflammation | day 7 after start of therapy
  Patients achieving 25% reduction in hyperinflammation score (CIS) compared to baseline at day 7

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hochhaus, Prof. Dr., Principal Investigator — University Hospital Jena
Locations (6):
- Germany (6):
  - SRH Wald-Klinikum Gera GmbH, Gera
  - University Hospital Jena, Jena
  - UKSH, Campus Lübeck, Lübeck
  - Klinikum der Landeshauptstadt Stuttgart gKöR, Stuttgart
  - Universitätsklinikum Ulm, Ulm
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen GmbH, Villingen-Schwenningen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hammersen J, Birndt S, Dohner K, Reuken P, Stallmach A, Sauerbrey P, La Rosee F, Pfirrmann M, Fabisch C, Weiss M, Trager K, Bremer H, Russo S, Illerhaus G, Dromann D, Schneider S, La Rosee P, Hochhaus A. The JAK1/2 inhibitor ruxolitinib in patients with COVID-19 triggered hyperinflammation: the RuxCoFlam trial. Leukemia. 2023 Sep;37(9):1879-1886. doi: 10.1038/s41375-023-01979-w. Epub 2023 Jul 28. PMID 37507425
- [Derived] La Rosee F, Bremer HC, Gehrke I, Kehr A, Hochhaus A, Birndt S, Fellhauer M, Henkes M, Kumle B, Russo SG, La Rosee P. The Janus kinase 1/2 inhibitor ruxolitinib in COVID-19 with severe systemic hyperinflammation. Leukemia. 2020 Jul;34(7):1805-1815. doi: 10.1038/s41375-020-0891-0. Epub 2020 Jun 9. PMID 32518419